CLINICAL TRIAL: NCT00530998
Title: Natural Orifice Translumenal Endoscopic Surgery (NOTES): Laparoscopic Assisted Trans-Vaginal Appendectomy and Cholecystectomy
Brief Title: Minimally Invasive Surgery: Using Natural Orfices
Acronym: NOTES
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Santiago Horgan, Professor of Surgery, University of California, San Diego
Other Study IDs: 071115, 140015
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Appendicitis; Cholelithiasis; Gallstones
Keywords: appendicitis; cholelithiasis; Gallstones
MeSH Terms: conditions — Appendicitis; Cholelithiasis; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Group #1 NOTES Appendectomy - Transvaginal approach
  Interventions: Procedure: Transvaginal Appendectomy
- 2: Group #2 NOTES Cholecystectomy - Transvaginal approach
  Interventions: Procedure: Transvaginal Cholecystectomy

INTERVENTIONS:
Procedure: Transvaginal Appendectomy — The appendix will be removed via an incision in the vagina.
  Groups: 1
Procedure: Transvaginal Cholecystectomy — The gallbladder will be removed via an incision in the vagina.
  Groups: 2

SUMMARY:
This is an observational study of pain and outcomes from females undergoing transvaginal NOTES removal of their appendix or gallbladder. Female subjects who elect to have a transvaginal NOTES removal of their appendix or gallbladder and agree to be in this study (through signature on the informed consent form) will be followed per standard of care, with additional follow-up for data collection including the following:

* Subjects will complete a 7 day pain/temperature log after surgery
* Subjects will complete a standardized sexual function questionnaire (Female Sexual Function Index) prior to surgery and 6 months after surgery
* Subjects will receive a phone call at 6 months and at 1 year after surgery to capture data related to safety, adverse events, hospitalizations and patient satisfaction

Additional data related to pain and outcomes will be collected at baseline/screening and at follow-up as necessary.

ELIGIBILITY:
Inclusion criteria for transvaginal appendectomy:

1. Females between the ages of 18-75
2. Clinical diagnosis of appendicitis
3. Emergency room evaluation within 36 hours of the onset of pain
4. ASA Classification 1
5. Mentally competent to give informed consent
6. Scheduled to undergo a transvaginal NOTES appendectomy.

Exclusion criteria for transvaginal appendectomy:

1. Pregnant women (need to have negative icon in ER)
2. Morbidly obese patients (BMI >35)
3. Patients who are taking immunosuppressive medications or are immunocompromised
4. Patients with evidence of an abdominal abscess or mass
5. Patients who present with a clinical diagnosis of sepsis or peritonitis
6. Patients who have a history of prior transvaginal surgery. Patients with prior laparoscopic surgery will be included.
7. Patients who endorse a history of ectopic pregnancy, pelvic inflammatory disease (PID), or severe endometriosis
8. Patients with diffuse peritonitis on clinical exam
9. Patients on blood thinners or aspirin or abnormal blood coagulation tests

Inclusion criteria for transvaginal cholecystectomy:

1. Females between the ages of 18 and 75
2. Diagnosis of gallstone disease which requires cholecystectomy
3. ASA class 1
4. Mentally competent to give informed consent
5. Scheduled to undergo a transvaginal NOTES cholecystectomy

Exclusion criteria for transvaginal cholecystectomy:

1. Pregnant women
2. Morbidly obese patients (BMI > 35)
3. Patients who are taking immunosuppressive medications and/or immunocompromised
4. Patients with severe medical comorbidities will be excluded.
5. Patients with a presumed gallbladder polyps, mass or tumor
6. Patients with a history of prior transvaginal surgery. Patients with prior laparoscopic surgery will be included.
7. Patients with a history of ectopic pregnancy, pelvic inflammatory disease, or severe endometriosis
8. Patients with known common bile duct stones
9. Patients on blood thinners or aspirin or abnormal blood coagulation tests

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group #1: NOTES Appendectomy - Transvaginal approach:
  Subjects will be female between the ages of 18-75 who present to the emergency room and are subsequently diagnosed with acute appendicitis. Following diagnosis, investigators will determine if the procedure can be completed via the transvaginal approach. If the patient satisfies the listed criteria then researchers will present study information and offer participation.
  Group # 2: NOTES Cholecystectomy - Transvaginal approach:
  Female subjects, between the ages of 18-75 who present in the UCSD surgery clinic for elective cholecystectomy will be offered participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-09; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of transvaginal NOTES appendectomies and cholecystectomies (through data collection). | 1 year

SECONDARY OUTCOMES:
To evaluate pain associated with the transvaginal approach (through data collection). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Horgan, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States